CLINICAL TRIAL: NCT00252213
Title: B-Type Natriuretic Peptide (Nesiritide) and Post Myocardial Infarction Left Ventricular Remodeling: Pilot Study Assessing Safety
Brief Title: BELIEVE Study: Nesiritide and Post Myocardial Infarction Left Ventricular Modeling
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: recruitment of subjects was halted prematurely. recruiting subjects halted prematurely
Sponsor: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1218-02; I704.358
Record Dates: First submitted 2005-11-10; First posted 2005-11-11 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-12

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

INTERVENTIONS:
Drug: Human BNP

SUMMARY:
This study is being done to determine the effects (good and bad) of intravenous infusion of a human brain natriuretic peptide (BNP), Natrecor (nesiritide), a hormone produced by the heart in persons who have just suffered a heart attack. The human BNP, Natrecor (nesiritide) has been approved by the United States Food and Drug Administration (FDA) to be given intravenously for the management of acute heart failure. It is unknown if human BNP may have good effects on the pumping function of the heart after a heart attack.

DETAILED DESCRIPTION:
During the 72 hours of intravenous (IV) nesiritide infusion, if the systolic blood pressure decreases to less than 90 mmHg for 5 minutes, the coronary care unit (CCU) sx will be notified and if the systolic blood pressure has not increased to > or equal to 90 mmHg within 45 minutes, the nesiritide infusion will be stopped. All patients will receive other medical therapy as determined appropriate by the physician except for angiotensin converting enzyme inhibitor (ACEI), which will be started 24 hours after IV nesiritide. Lisinopril will be started 24 hours after the start of IV nesiritide at an initial dose of 2.5 mg and to be titrated up by the participants' physician according to their clinical status. The window for the lisinopril doses would be +/- 1 hour.

Patients with any signs or symptoms of post revascularization ischemia will be discontinued from the study.

Blood for the measurement of renin, angiotensin II (Ang II), aldosterone (Aldo), endothelin (ET)-1, norepinephrine, atrial natriuretic peptide (ANP), brain natriuretic peptide (BNP), cGMP, C reactive protein, tumor necrosis factor (TNF)-alpha, matrix metalloproteinase (MMP)-2 and tissue inhibitor of metalloproteinase (TIMP)-2 will be drawn before the initiation of IV nesiritide, six hours into the infusion before the initiation of ACEI and just before completion of the 72 hour infusion. The window for the blood draw for the six hour time point would be +/- 1 hour and the 72 hour time point would be +/-1 hour or just prior to discharge but not less than 66 hours.

MUGA will be performed within 24 hours after the initiation of the IV nesiritide to assess systolic and diastolic volumes and LV ejection fraction (EF).

Follow up at 4 weeks:

All patients, whether they complete the entire 72 hours of the nesiritide infusion or not, will return 1 month later for a repeat MUGA and blood draw for the neurohumoral profiling and pregnancy test if required by nuclear cardiology. The visit window for the one month return would be 30 to 40 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ST elevation myocardial infarction of at least > 2mV ST elevation in two or more anterior precordial leads, with successful revascularization (Thrombolysis in Myocardial Infarction [TIMI] grade 3 flow) of the lesion within 24 hours of chest pain as documented by coronary angiogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2002-08; Study Completion 2006-01

PRIMARY OUTCOMES:
Determine the safety of nesiritide at two different dose levels of 0.003 µg/Kg/min and 0.006 µg/Kg/min focusing on the occurrence of hypotension (yes versus no)
Dosing finding comparing the efficacy of 0.003 µg/Kg/min and 0.006 µg/Kg/min on the suppression of aldosterone at 6 hours after the start of infusion as compared to baseline, as a marker of the neurohumoral activity of BNP

SECONDARY OUTCOMES:
Compare the safety of the two doses on left ventricular (LV) remodeling by determining the LV volume and function by multiple gate acquistion scan (MUGA)

CONTACTS AND LOCATIONS:
Overall Officials: Horng H. Chen, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States